CLINICAL TRIAL: NCT07298408
Title: Cannabidiol for the Treatment of Diabetic Peripheral Neuropathy: Pilot Study
Acronym: CBD-DPN1
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Florida A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TMH2025-3; 175348 (Other: U.S. Food and Drug Administration)
Record Dates: First submitted 2025-12-19; First posted 2025-12-23 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Peripheral Neuropathic Pain (DPN); Diabetic Neuropathies
Keywords: Placebo; Pain Management; Quality of Life; Cross-Over Studies; Double-Blinded Placebo Contolled; Cannabidiol
MeSH Terms: conditions — Diabetic Neuropathies; Agnosia | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: 1. CBD Isolate Phase 1 Placebo Phase 2
  2. CBD Isolate Phase 2 Placebo Phase 1
  3. CBD Full-spectrum Phase 1 Placebo Phase 2
  4. CBD Full-spectrum Phase 2 Placebo Phase 1
  There is a two-weeks washout period between the two phases of the study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1. CBD Isolate Phase 1 (Placebo Phase 2) (Experimental): Participants randomized to Arm 1 will be given CBD Isolate tincture 100 mg/ml (50 mg twice daily for a total of 100 mg daily) for 6 weeks in Phase 1. After a 2-week washout period they will be given an identical appearing placebo tincture for an additional 6 weeks. The bottles will be labeled: "TMH CBD for DPN Trial: (number) A" and "TMH CBD for DPN Trial: (number)B", where A refers to the vials to be used in phase one and B to the vials used for phase two. Since a vial contains a 30-day supply and each phase lasts 42 days, the participants will receive two identically labelled vials at the beginning of each phase.1
  Interventions: Drug: Cannabidiol (CBD) oral solution
- 2. Placebo Phase 1 (CBD Isolate Phase 2) (Placebo Comparator): Participants randomized to Arm 2 will be given a placebo tincture (0.5 ml twice daily for a total of 1 ml daily) for 6 weeks in Phase 1. After a 2-week washout period, they will be given the active tincture containing 100 mg of CBD isolate (100 mg/ ml) to use 0.5 ml twice daily for an additional 6 weeks. The bottles will be labeled: "TMH CBD for DPN Trial: (number) A" and "TMH CBD for DPN Trial: (number)B", where A refers to the vials to be used in phase one and B to the vials used for phase two. Since a vial contains a 30-day supply and each phase lasts 42 days, the participants will receive two identically labelled vials at the beginning of each phase.
  Interventions: Drug: Placebo in MCT oil oral solution
- 3. CBD Full-spectrum Phase 1 (Placebo Phase 2) (Experimental): Participants randomized to Arm 3 will be given a Full-spectrum CBD isolate tincture with 100 mg of hemp-derived CBD isolate /ml (using 0.5 ml; 50 mg twice daily for a total of 100 mg daily) for 6 weeks in Phase 1. After a 2-week washout period they will be given an identical appearing placebo tincture for an additional 6 weeks. The bottles will be labeled: "TMH CBD for DPN Trial: (number) A" and "TMH CBD for DPN Trial: (number)B", where A refers to the vials to be used in phase one and B to the vials used for phase two. Since a vial contains a 30-day supply and each phase lasts 42 days, the participants will receive two identically labelled vials at the beginning of each phase.
  Interventions: Drug: Full-Spectrum CBD hemp extract oral solution
- 4. Placebo Phase 1 (CBD Full-spectrum Phase 2) (Placebo Comparator): Participants randomized to Arm 4 will be given a placebo tincture (0.5 ml twice daily for a total of 1 ml daily) for 6 weeks in Phase 1. After a 2-week washout period, they will be given the active tincture containing 100 mg of CBD Full-spectrum isolate (100 mg/ ml) to use 0.5 ml twice daily for an additional 6 weeks. The bottles will be labeled: "TMH CBD for DPN Trial: (number) A" and "TMH CBD for DPN Trial: (number)B", where A refers to the vials to be used in phase one and B to the vials used for phase two. Since a vial contains a 30-day supply and each phase lasts 42 days, the participants will receive two identically labelled vials at the beginning of each phase.
  Interventions: Drug: Placebo in MCT oil oral solution

INTERVENTIONS:
Drug: Cannabidiol (CBD) oral solution — Strawberry-flavored Cannabidiol oral solution in medium-chain triglyceride (MCT) oil, administered orally, 100mg/ml in a 30 ml dropper bottle.
  Arms: 1. CBD Isolate Phase 1 (Placebo Phase 2)
Drug: Full-Spectrum CBD hemp extract oral solution — Strawberry-flavored Full-Spectum Cannabidiol oral solution in medium-chain triglyceride (MCT) oil, administered orally, 100mg/ml in a 30 ml dropper bottle.
  Arms: 3. CBD Full-spectrum Phase 1 (Placebo Phase 2)
Drug: Placebo in MCT oil oral solution — Strawberry-flavored medium-chain triglyceride (MCT) oil, administered orally, 30 ml dropper bottle.
  Arms: 2. Placebo Phase 1 (CBD Isolate Phase 2); 4. Placebo Phase 1 (CBD Full-spectrum Phase 2)

SUMMARY:
The "Cannabidiol for the Treatment of Diabetic Peripheral Neuropathy: Pilot study (CBD-DPN1)" is a double-blinded, placebo-controlled, crossover pilot study evaluating the efficacy of Cannabidiol (CBD) and full-spectrum CBD (fsCBD) tinctures in treating Diabetic Peripheral Neuropathy (DPN)-associated pain. DPN is a common, highly distressing complication of diabetes, characterized by chronic pain and loss of sensory function, for which currently available treatments primarily offer only symptomatic relief. CBD and fsCBD are being investigated for their potential neuroprotective and analgesic effects by regulating inflammation and oxidative stress.

The study aims to recruit 12 to 20 adult participants who have mild to moderate DPN. Subjects will receive either an active treatment (CBD isolate or fsCBD in MCT oil, dosed at 50 mg twice daily for a total of 100 mg daily) or a placebo during two sequential 6-week phases. The overall objective of this pilot phase is primarily methodological: to test and refine the clinical protocol, assess patient compliance and acceptability of the CBD formulations, and generate sufficient data to calculate the necessary sample size for a larger, definitive study. Efficacy will be measured using objective and subjective metrics, including DPN severity (DN4 Assessment Tool and DPNCheck™ for nerve conduction velocity) and pain level (PainDetect Questionnaire). Secondary outcomes include evaluating mood (HADS), sleep quality (MOS Sleep Scale), and quality of life (EQ-5D-5L).

DETAILED DESCRIPTION:
The Cannabidiol for the Treatment of Diabetic Peripheral Neuropathy: Pilot study (CBD-DPN1) is an interventional, double-blinded, placebo-controlled, crossover pilot study investigating the efficacy of cannabidiol (CBD) formulations in treating diabetic peripheral neuropathy (DPN)-associated pain. This study operates under an Investigational New Drug (IND) application cleared by the U.S. Food and Drug Administration (FDA).

Scientific Rationale and Objectives DPN is a widespread and highly distressing complication of Type 2 Diabetes (T2D), leading to chronic pain, numbness, and significant loss of quality of life. Current treatments primarily offer symptomatic relief without halting the disease progression. CBD is a non-psychoactive phytocannabinoid attracting attention for its neuroprotective action and potential therapeutic effect against DPN pain. Mechanistically, CBD is hypothesized to reduce neuropathic and musculoskeletal pain by regulating inflammation and oxidative stress through antagonism of CB1 receptors, agonism of CB2 receptors, and modulation of TRPV1 ion channels. Preclinical data further suggests CBD significantly improves behavioral DPN parameters in diabetic rat models and positively regulates mitochondrial homeostasis pathways (Nrf2-SIRT1 axis) in Schwann cells.

The overall objective is to determine the efficacy of CBD and Full-spectrum CBD delivered as a tincture in treating DPN-associated pain. As a pilot study, the primary objectives are methodological: to evaluate and refine the clinical protocol, assess patient compliance and acceptability of the CBD formulations, test organoleptic acceptability (if participants can discern active agent from placebo), and gather initial data necessary for power size estimates for a future large-scale study.

Study Design and Treatment Protocol The study targets the recruitment of approximately 30 subjects for screening, with a goal of enrolling a minimum of 12 to 20 adults with mild to moderate DPN. The total duration for each participant is about 4 months.

Crossover Design and Blinding: Participants are randomized into four treatment sequences, ensuring each subject receives both an active treatment phase and a placebo phase across the two sequential 6-week treatment periods (Phase I and Phase II). This design ensures that following the enrollment of 4, 8, 12, 16, or 20 participants, there is an equal distribution of subjects across the four treatment combinations. The study is double-blinded, meaning neither the subject nor the clinical investigators will know the assignment of the active agent or placebo during either phase.

Interventional Agents and Dosing: The investigational products are administered orally in Medium-Chain Triglyceride (MCT) oil:

1. CBD Isolate Tincture: Pure Cannabidiol isolate in MCT oil. The formulation is a high concentration oral solution of CBD (100 mg/mL), provided by the manufacturer Sunflora.
2. Full-spectrum CBD (fsCBD) Tincture: Cannabidiol hemp extract in MCT oil, containing 85.75 mg of CBD and approximately 13 mg of other cannabinoids (like CBG, CBN, and CBC) per milliliter, and less than 0.3% THC.
3. Placebo: MCT oil formulated identically with natural strawberry flavoring to match the active agents, helping to maintain blinding.

The dose of the active agent (CBD or fsCBD) is 100 mg daily. This daily dose is split, requiring subjects to take 0.5 ml (50 mg) twice daily with a meal (breakfast and supper) to optimize absorption. This dose is relatively low, being less than 2 mg/kg for most participants, which is several-fold lower than doses associated with statistically significant adverse effects observed in epilepsy trials (10-20 mg/kg).

Assessments and Schedule Outline The study involves clinic visits at Day 0, Day 7 (Start of Phase I), Day 49 (End of Phase I/Start of Phase II), and Day 91 (End of Phase II), followed by a phone follow-up at Day 105.

* Objective Neuropathy Measurement: The degree of peripheral neuropathy and the progression of the disease is monitored using a needleless, validated, point-of-care Nerve Conduction Test (NCT) performed with the DPNCheck™ instrument. NCV/SNAP amplitude testing is conducted at baseline (Day 0), mid-study (Day 49), and end-of-study (Day 91). A brief physical exam, including testing for hypoesthesia and allodynia using a nylon filament and a brush, is conducted at baseline and end of phase visits.
* Subjective Metrics: Multiple validated instruments are used to assess DPN symptoms, mood, and quality of life:

  * Pain: PainDetect Questionnaire (slightly modified to quantify changes) to assess allodynia and hyperalgesia.
  * Sleep: MOS Sleep Scale.
  * Mood/Anxiety: Hospital Anxiety and Depression Scale (HADS).
  * Quality of Life: EQ-5D-5L Quality of Life Scale.
  * Subjects are trained to complete these questionnaires at Day 7 under supervision and subsequently complete them at home every two weeks.
* Compliance: Compliance is objectively assessed by measuring the volume of remaining oil in the vials returned by the subject at the end of Phases I (Day 49) and II (Day 91), and by scoring the completeness of the questionnaires. Subjects are also debriefed at the final visit regarding their perception of the active vs. placebo phases.

Safety Management and Withdrawals Given the low anticipated toxicity profile of the low CBD dose, a formal Data Safety Monitoring Board (DSMB) is not warranted for this pilot study; oversight is managed closely by the Principal Investigators (PIs).

* Liver Function Monitoring: Because CBD can interact with cytochrome P450 enzymes (e.g., CYP3A4, CYP2C9) and high doses have been linked to liver enzyme elevations, liver function tests (ALT and AST) are checked before the start of the trial (or current results reviewed) and again at the end of treatment (Day 91). Subjects with severe active liver disease are excluded, although those with Non-Alcoholic Fatty Liver Disease (NAFLD) with only mildly elevated enzymes (ALT or AST the ULN) are permitted due to the high prevalence of NAFLD in the target T2D population.
* Drug-Drug Interactions (DDIs): Patients currently using medications metabolized by key CYP450 enzymes (such as Warfarin, Amiodarone, Cyclosporine, and certain anticonvulsants) are excluded to mitigate the risk of DDIs, as CBD can reduce the activity of these metabolizing enzymes.
* Stopping Criteria: Treatment will be immediately discontinued for any participant exhibiting worsening cardiovascular symptoms (e.g., hypotension, tachycardia, syncope, worsening hypertension) or neuropsychiatric symptoms (anxiety, paranoia). Participants are withdrawn for non-compliance, new exclusion criteria (such as pregnancy), or any adverse event severe enough to require hospitalization and reasonably attributed to the treatment.

The DPNCheck™ instrument performs a needleless nerve conduction test, which involves placing electrodes on the skin and running a small current, minimizing risks of infection or injury associated with venipuncture. Subjects are instructed on side effects of the interventional agents , which are generally expected to be mild and self-limiting, such as drowsiness, diarrhea, or dry mouth.

ELIGIBILITY:
Inclusion Criteria

1. Adult aged 40 to 70 years
2. Diagnosis of Type 2 Diabetes
3. Ambulatory and independently living adult
4. Minimum body weight of 50 kg (to ensure daily dose ≤2 mg/kg)
5. Physical exam completed within the previous 6 months
6. Liver Function Studies (ALT and AST) completed within the previous six months showing normal values
7. If NAFLD is present, ALT and AST levels are ≤2 times the Upper Limit of Normal (ULN)
8. DN4 questionnaire results indicate mild to moderate DPN
9. Nerve Conduction Test (NCT) confirms at least mild DPN
10. Signed ICF/Screening Consent
11. Able to complete required questionnaires (adequate vision)

Exclusion Criteria:

1. High-risk or severely ill individuals (e.g., high risk for general anesthesia, significant limitations due to heart/lung disease, ascites, renal failure, loss of limbs from diabetic complications)
2. Uncontrolled or severe cardiovascular disease (e.g., unstable angina, uncontrolled heart failure, recent myocardial infarction)
3. History of atrial fibrillation, dysrhythmias, MI within the previous 2 years, or stroke
4. Severe respiratory illness (e.g., uncontrolled asthma, COPD with frequent exacerbations, oxygen dependence)
5. Severe or uncontrolled liver disease (e.g., cirrhosis, active viral hepatitis A, B, or C, autoimmune hepatitis, uncontrolled primary biliary cholangitis or primary sclerosing cholangitis)
6. Elevation of liver enzymes (ALT or AST) exceeding 2 times the ULN, or bilirubin exceeding the ULN
7. Severe or uncontrolled kidney disease (e.g., end-stage renal disease requiring dialysis, uncontrolled nephrotic syndrome)
8. History of malignancy within the past 5 years (excluding certain low-risk non-melanoma skin cancers)
9. History of a seizure disorder
10. Blindness (poor vision preventing questionnaire completion)
11. Known allergy or previous adverse reaction to any ingredient, including natural strawberry flavoring
12. Reproductive Health (Women Only)
13. Currently pregnant or lactating
14. Women who can get pregnant who are not using acceptable methods of birth control
15. Current uncontrolled mental health conditions (e.g., major depressive episode with active suicidal ideation, bipolar disorder with current manic/hypomanic episode, or psychosis)
16. Diagnosis of a major depressive episode with active suicidal ideation and/or a plan to attempt suicide within the previous 5 years
17. Attempted suicide in the last 10 years
18. C-SSRS Suicide Ideation Subscore ≥5 at study onset
19. HADS-D score ≥15 at study onset
20. Used cannabis products in the past 30 days
21. Current use or history of illicit drug use or misuse of prescription medications within the previous 5 years
22. Heavy drinking (≥8 drinks/week for women; ≥15 drinks/week for men)
23. Taking medications that are known to cross-reacting with CBD or Cannabiods

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
DPN Pain Level | Baseline (Day 0), Day 7, Day 21 (at home by subject), Day 35 (at home by subject), End of Phase I (Day 49), Day 63 (at home by subject), Day 77 (at home by subject), End of Phase II (Day 105).
  Pain level will be assessed using the slightly modified "PainDETECT" Questionnaire. This instrument rates subjective pain 0 - 10 (zero no pain, 10 the worst) for current, average and worst over the last 4 weeks. It additionally scores neuropathic symptoms on a scale of zero to 35, with zero being no symptoms to 35 being the worst.
Diabetic peripheral neuropathy diagnosis | Baseline Screening (Day 0)
  DPN severity will be assessed using the DN4 Assessment Tool (including a clinical assessment of hypoesthesia and allodynia). The DN4 tool consists of 10 items across four sections, including both patient interview questions and a physical examination. Each "yes" answer receives 1 point, and each "no" answer receives 0 points. The points from all 10 items are summed to get a total score ranging from a minimum of 0 to a maximum of 10. A total score of 4 or more (≥4) suggests the presence of neuropathic pain. A score of 3 or below indicates that neuropathic pain is unlikely. A higher score is associated with worse DPN.
Diabetic Neuropathy Severity | Baseline, End of Phase I (Day 49) (for NCT), End of Phase II (Day 91) (for NCT).
  The DPNCheck™ instrument will be used to assess sural nerve conduction velocity (NCV) and sensory nerve action potential (SNAP) amplitude. Amplitude, The typical normal ranges are > 40 m/s for SNAV and > 4 µV SNAP, though values vary by study; lower values indicate worse neuropathy severity, with thresholds like \(<40\) m/s for SNCV and \(<5\) µV (or even \(<4\) µV) for SNAP signaling mild-to-moderate damage, while amplitudes below 1.5 µV may register as zero due to device limits. Device Limitation: Values below 1.5 µV may be registered as 0 µV. Mild DPN: May show delayed SNCV (< 40 m/s) or low amplitude. Moderate DPN: Often characterized by reduced SNAP amplitude (e.g., < 5 µV). Severe DPN: Significant decreases in both amplitude and velocity, with very low or undetectable signals

SECONDARY OUTCOMES:
Sleep Quality | Periodically over the approximately 4 month study duration
  Assessment of changes in sleep quality using the sleep scale from the "Medical Outcomes Study" (MOS). The instrument includes 10 Likert-type responses (1 - 6 scale) and are mostly reverse-scoring items (marked with 'R') to transform them into a 0-100 scale. Higher scores generally mean better sleep for "get enough sleep to feel rested" but higher scores indicate more problems for indices like Sleep Disturbance, with specific items like Sleep Quantity measured in hours. Final scores are often expressed as T-scores (mean 50, SD 10) for general population comparison. In the final score higher scores = better sleep
Mood and Depression | Periodically over the approximately 4 month study duration
  Assessment of changes in mood and depression using the Hospital Anxiety and Depression Scale (HADS) instrument.There are 14 Items and the scale has two sub-scales: Anxiety (A) and Depression (D). Each item is rated 0 (not at all) to 3 (definitely/very much). Scoring ranges from 0-7: Normal, 8-10: Borderline, abnormal/Mild, 11-14: Moderate, and 15-21: Severe. There are separate m measures for anxiety and depression. Thus, a higher score is worse.
Quality of Life Index | Periodically over the approximately 4-month study duration
  Assessment of changes in quality of life (using the EQ-5D-5L Quality of Life Scale). The EQ-5D-5L asks about five health dimensions (mobility, self-care, activities, pain/discomfort, anxiety/depression), each with 5 levels (1=no problems, 5=extreme). This is converted into a single "utility" score (0 to 1, with negative values possible) Higher scores are worse while score of 1 is having no problems in that dimension. The measure also includes a separate 0-100 Visual Analogue Scale (EQ-VAS) for self-rated health, with zero as the worst possible health imagined and 100 the best.
Patient Compliance | End of Phase I (Day 49) End of Phase II (Day 105)
  Assessed by measuring the remaining oil volume in the vials and scoring the completeness of the questionnaires. The higher the volume deviates from the prescribed use, the worse the compliance. The lower the percentage of questionnaires fully completed, the lower the compliance.
Liver Function Monitoring (Safety Measure) | Baseline, (if previous results are > 3 months old), End of Phase II (Day 105)
  Measurement of liver enzymes: Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) (Liver function tests - LFTs). Higher LFT values indicate worse liver injury. Volunteers with LFT greater than two times the upper reference value at baseline will be excluded from participation. If LFT levels rise to exceed two-times the upper reference value during the study, the study medication will be stopped.

CONTACTS AND LOCATIONS:
Locations (1):
- the FSU TMH Family Practice Residency Program, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared primarily with the Sponsor and their designated agents/collaborators for the purposes of study monitoring, data analysis, protocol evaluation, and generating initial data for power size estimates needed for a larger, definitive study. Regulatory agencies, including the Food and Drug Administration (FDA), may also inspect and copy the information.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be compiled and prepared for analysis following the completion of the trial and the final follow-up visit (Day 105). The sponsor will reveal the treatment labeling data after the trial for data analysis
Access Criteria: Access to the coded IPD will be limited to the study team, the Sponsor (Florida A&M University), and its agents or collaborators (e.g., the funder, Consortium for Medical Marijuana Clinical Outcomes Research (CCORC)) necessary for study conduct, oversight, and data analysis.